CLINICAL TRIAL: NCT02015481
Title: Multi-Center, Dose-Escalation Study, to Assess Safety, Tolerability and Efficacy of Intravenous Cabaletta® in OPMD Patients
Brief Title: Safety Tolerability and Efficacy Study of Cabaletta to Treat Oculopharyngeal Muscular Dystrophy (OPMD) Patients
Acronym: HOPEMD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bioblast Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBCO-001
Record Dates: First submitted 2013-12-08; First posted 2013-12-19 (Estimated); Results first posted 2017-08-23 (Actual); Last update posted 2017-10-17 (Actual); Status verified 2017-09

CONDITIONS: Oculopharyngeal Muscular Dystrophy
Keywords: Case control, safety, tolerability, efficacy.
MeSH Terms: conditions — Muscular Dystrophy, Oculopharyngeal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cabaletta 30gr. (Experimental): weekly IV of Cabaletta 30gr.
  Interventions: Drug: Cabaletta

INTERVENTIONS:
Drug: Cabaletta

SUMMARY:
The Purpose of this study is to assess the Safety, Tolerability and Efficacy of Intravenous Cabaletta® in Oculopharyngeal Muscular Dystrophy (OPMD) Patients.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* 18 - 80 years (inclusive) of age
* Clinically and genetically diagnosed as OPMD
* Moderate dysphagia (abnormal drinking test at screening and on the first dosing day, before drug administration)
* Patients who provide written informed consent to participate in the study
* Body Mass Index (BMI) <30 kg/m2

Exclusion Criteria:

* Diabetes mellitus type 1 or 2
* Other major diseases, e.g.: renal failure (creatinine clearance <60ml/min), liver failure and chronic liver diseases (e.g. hepatitis B or C) , HIV carriers, tuberculosis, SLE, rheumatoid polyarthritis, sarcoidosis, collagenosis
* Uncontrolled heart disease , CHF,
* Other neuromuscular diseases
* Other disorders associated with esophageal dysphagia: e.g. severe gastroesophageal reflux (GERD), esophageal stricture due to mechanical or chemical trauma, infection (e.g. esophageal moniliasis), drug-induced dysphagia (e.g. bisphosphonates), esophageal rings and webs, spastic motility disorders of the esophagus.
* History of malignancy (except non-invasive skin malignancy)
* History of neck irradiation
* Pregnant or currently lactating women
* Obesity (BMI≥ 30) and associated morbidity
* Prior pharyngeal myotomy
* Weight loss of more than 10% in the last 12 months.
* Known hypersensitivity to any ingredients in the injection
* Patient receiving anticoagulant treatment (e.g. warfarin)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoseph Caraco, M.D, Principal Investigator — Hadassah Medical Organization; Bernard Brais, MD, Principal Investigator — McGill University
Locations (4):
- United States (2):
  - UCLA, Los Angeles, California
  - Tahseen Mozaffar, Orange, California
- Montreal Neurological Institute, McGill University, Montreal, Quebec, Canada
- Hadassah medical center, Jerusalem, Israel

RESULTS

PARTICIPANT FLOW:
Groups:
- Cabaletta 30gr: weekly IV of Cabaletta 30gr
  Cabaletta
Period: Overall Study
Arm/Group | Cabaletta 30gr
Started | 25
Completed | 24
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Groups:
- Cabaletta 30gr.: weekly IV of Cabaletta 30gr.
  Cabaletta
Arm/Group | Cabaletta 30gr.
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (8.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 12
Region of Enrollment [Number; unit: participants]
  Canada | 11
  Israel | 14

OUTCOME MEASURES:

1. Primary Outcome: Safety Lab Evaluations
Description: Change from baseline in safety labs including hematology, coagulation, chemistry, renal function, and liver function tests at week 24 .
Time Frame: 24 weeks
Population: 24 patients were available for analysis at week 24. Not all patients had all labs performed. Missing data accounts for the differing number of patients with specific lab values.
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Cabaletta 30gr.
Number analyzed (Participants) | 24
percentage change from baseline
  White Blood Cell Count | -4.0 (16.69)
  Red Blood Cell Count: number analyzed (Participants) | 13
  Red Blood Cell Count | 0.1 (0.42)
  Hemoglobin: number analyzed (Participants) | 13
  Hemoglobin | 0.2 (7.98)
  Hematocrit: number analyzed (Participants) | 13
  Hematocrit | 1.1 (9.28)
  Platelets | -0.5 (13.42)
  Alanine Aminotransferase | -0.8 (34.59)
  Aspartate Aminotransferase: number analyzed (Participants) | 23
  Aspartate Aminotransferase | -5.7 (30.93)
  Creatinine phosphokinase | 6.8 (37.12)
  Gamma-Glutamyl Transferase: number analyzed (Participants) | 23
  Gamma-Glutamyl Transferase | 9.3 (28.73)
  Total Bilirubin: number analyzed (Participants) | 13
  Total Bilirubin | 37.2 (46.02)
  Glucose: number analyzed (Participants) | 13
  Glucose | 12 (15.93)
  Lactose Dehydrogenase: number analyzed (Participants) | 23
  Lactose Dehydrogenase | 23 (0.9)
  Prothrombin Time: number analyzed (Participants) | 22
  Prothrombin Time | 7.1 (12.62)
  International Normalized Ratio: number analyzed (Participants) | 22
  International Normalized Ratio | 1.3 (8.48)

2. Secondary Outcome: Drinking Test Score
Description: Change from baseline in ice water drinking time, in seconds, at week 24. Times greater than 8 seconds to complete the drinking test are considered abnormal.
Time Frame: 24 weeks
Population: 22 patients had data available for analysis at week 24
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Cabaletta 30gr
Number analyzed (Participants) | 22
percentage change from baseline | -33.8 (34.89)

3. Secondary Outcome: Videofluoroscopy (VFS) Score
Description: Penetration aspiration score results assessed by VFS comparing baseline, prior to treatment, to week 24. This is an 8 point scale. The higher the number the greater the risk of aspiration. The result reported is the difference from the baseline scores.
Time Frame: 24 Weeks
Population: 11 patients had valid baseline data and week 24 data
Measure: Mean (Standard Deviation); unit: Points on an 8 point scale
Arm/Group | Cabaletta 30gr
Number analyzed (Participants) | 11
Points on an 8 point scale | 0.1 (1.27)

4. Secondary Outcome: SWAL-QOL, Swallowing Quality of Life Questionnaire
Description: Summary of Quality of Life in Swallowing Disorders total symptom score results over time, change from baseline at weeks 12 and 24 This is a 100 point scale. The higher the number the better the quality of life.
Time Frame: 28 weeks
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Cabaletta 30gr
Number analyzed (Participants) | 24
percentage change from baseline | 12.4 (16.87)

ADVERSE EVENTS:
Time Frame: 28 weeks
Arm/Group | Cabaletta 30gr
All-Cause Mortality (participants affected / at risk) | 1/25
Serious Adverse Events (participants affected / at risk) | 2/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabaletta 30gr (N=25)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabaletta 30gr (N=25)
Abdominal Pain (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Toothache (Gastrointestinal disorders) | 2 (2)
Administrative Site Bruise (General disorders) | 4 (5)
Asthenia (General disorders) | 2 (2)
Fatigue (General disorders) | 4 (5)
Influenza Like Illness (General disorders) | 3 (3)
Pyrexia (General disorders) | 2 (2)
Bacteriuria (Infections and infestations) | 2 (3)
Nasopharyngitis (Infections and infestations) | 4 (5)
Pharyngitis (Infections and infestations) | 2 (3)
Urinary Tract Infection (Infections and infestations) | 3 (4)
Procedural Pain (Injury, poisoning and procedural complications) | 10 (14)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 7 (10)
Muscle Fatigue (Musculoskeletal and connective tissue disorders) | 3 (4)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Headache (Nervous system disorders) | 5 (10)
Elevated Urine Glucose Levels (Renal and urinary disorders) | 13 (35)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes